CLINICAL TRIAL: NCT01344499
Title: Clearance Rate of Peritoneal Fluid Assessed by Post-operative Ultrasound Decreases After Full Conditioning Pneumoperitoneum
Brief Title: Clearance Rate of Peritoneal Fluid After Full Conditioning Pneumoperitoneum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Jasper Verguts, MD, PhD, University Hospital, Gasthuisberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S52808
Record Dates: First submitted 2011-04-21; First posted 2011-04-29 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Laparoscopic Hysterectomy
Keywords: women; laparoscopic subtotal hysterectomy
MeSH Terms: interventions — Carbon Dioxide; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adept (Experimental): 1000ml Adept will be left in the abdomen and measured over time
  Interventions: Procedure: Carbon dioxide; Procedure: full conditioning; Drug: Adept
- Ringer-lactate (Active Comparator): 1000 ml of Ringer lactate left in the abdomen and measured over time
  Interventions: Procedure: Carbon dioxide; Procedure: full conditioning; Drug: Ringer Lactate

INTERVENTIONS:
Procedure: Carbon dioxide — standard pneumoperitoneum with 100% CO2
Procedure: full conditioning — Pneumoperitoneum with CO2 + 4% of oxygen + 10% nitrous oxide + 100% RH + T° 32°C
Drug: Adept — instillation of 1 liter of fluid at the end of laparoscopy
  Arms: Adept
Drug: Ringer Lactate — instillation of 1 liter of fluid at the end of laparoscopy
  Arms: Ringer-lactate

SUMMARY:
Measurement of residual peritoneal fluid after laparoscopic surgery

DETAILED DESCRIPTION:
Primary endpoints

* to evaluate whether the clearance rate of peritoneal fluid is exponential or linear over time. (absorption rate expected for Adept ~30-60 ml/h)
* to evaluate the role of the mesothelial barrier in this clearance rate.

Knowing that diffusion to and from peritoneal fluid decreases with increasing molecular weight (MW), our hypothesis is that clearance rate will decrease following peritoneal conditioning. Indeed a decreased mesothelial trauma (either through hypoxia or through denudation) and retraction will expose less the basal membrane

Secondary endpoints:

-To confirm the decrease in post-operative pain as measured by VAS-score and inflammation as measured by CRP and leucocytosis with the full conditioning of the pneumoperitoneum.

ELIGIBILITY:
Inclusion Criteria:

* Women planned to undergo a total or subtotal laparoscopic hysterectomy and having signed the informed consent.
* No limitation in body mass index or uterine size is made.

Exclusion Criteria:

* pregnancy
* immunodeficiency
* refuse or unable to sign informed consent
* chronic disease (i.e. COPD, Crohn, cardiac…)
* known allergy for Adept©

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
clearance rate of peritoneal fluid | 3 days after surgery
  We will estimate the residual volume of fluid in the abdominal cavity in a 30° anti-Trendelenburg position after 1 minute in this position. Measurements will be repeated daily until discharge.

SECONDARY OUTCOMES:
Pain and inflammation score | 3 days after surgery
  Postoperative pain will be assessed by the intake of ibuprofen or other pain killers and by Visual Analog Scale (VAS). Patients will be asked to locate their pain-symptoms (shoulder, subcostal, trocar wound and visceral pain) and score the severity. VAS will be collected 2-4 hours after surgery and every post-operative day until discharge.
  Daily routine blood samples will be obtained and CRP will be measured. Routinely time of first flatus or stools will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: JAsper Verguts, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, campus Gasthuisberg, Leuven, Belgium